CLINICAL TRIAL: NCT05052905
Title: Virtual Reality Based Rehabilitation of Vestibular and Oculomotor Function for Pediatric ABI in a Home Setting
Brief Title: VR-based Remote Rehabilitation for Pediatric ABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Libra At Home LTD (Industry)
Collaborators: Alyn Pediatric & Adolescent Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 041-21
Record Dates: First submitted 2021-08-25; First posted 2021-09-22 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Acquired Brain Injury
Keywords: Pediatric
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study (Experimental): Exercises
  Interventions: Device: LibraVR

INTERVENTIONS:
Device: LibraVR — LibraVR is a standalone VR-based rehabilitation software for use in physiotherapy. It is designed to work with standard off-the-shelf hardware that is tested and approved for use in conjunction with the software.
  LibraVR system consists of the software (LibraVR Clinic) running on a PC (database of patients, creation of protocols, uploading protocols to mobile), and the LibraVR Mobile APP that runs on commercial mobile smartphones embedded in a lightweight cardboard or plastic VR viewer that the child wears as they would eyeglasses. The software displays a range of immersive VR exercises.

SUMMARY:
The primary objective of this study is to evaluate the feasibility and effectiveness of an at-home program of VR-based vestibular and oculomotor rehabilitation on improving postural stability, ocular motility and activities of daily living for children with mild to severe ABI

ELIGIBILITY:
Inclusion Criteria:

* They are ALYN patients undergoing physiotherapy for mild to severe ABI;
* They experience symptoms of vestibular function such as vertigo, postural instability, or impaired ocular motility;
* They are between the ages of 8 and 18;
* The time since injury/event is between 10 days and 1 year after the injury/event;
* They are able to maintain stable and dynamic positioning of the head;
* They able to walk with or without assistive equipment, or use a wheelchairs with no need for head support, defined by a LSS (level of sitting scale) score of 3 or greater (scale range: 1-8);
* Are able to understand basic instructions;
* Have sufficient visual acuity and visual field to identify and track mid-size objects on a screen.

Exclusion Criteria:

* Psychological, neurological or cognitive disorders which could impede participation, such as a history of epileptic seizures;
* Untreated benign paroxysmal positional vertigo (BPPV);
* Are in early post-operative stages (to avoid risk of bleeding or cerebrospinal fluid leak);
* Hearing impairment.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Vestibular Oculomotor Motor Screening (VOMS) | 6 months
  Symptoms scoring from 0 (none) to 10 (severe)
Pediatric Vestibular Symptom Questionnaire (PVSQ) | 6 months
  Score ranging from 0 (never) to 33 (most of the time) with a 4-Likert scale
Convergence Insufficiency Symptom Survey (CISS) | 6 months
  Score ranging from 0 (never) to 56 (Always) with a 5-Likert scale
Dizziness Handicap Inventory (DHI) | 6 months
  Score ranging from 0 (none) to 100 (severe) with a 3-Likert scale
Dizziness Handicap Inventory for patients caregivers (DHI-PC) | 6 months
  Score ranging from 0 (none) to 100 (severe) with a 3-Likert scale
Pediatric Quality of Life Inventory (PEDSQL) | 6 months
  Score ranging from 0 (worst) to 100 (best) with a 5-Likert scale
Modified Clinical Test of Sensory Interaction in Balance (mCTSIB) | 6 months
  Time score ranging from 0 (unable to complete) to 120 (completed successfully) in one of three 30-seconds trials and four conditions
Berg Balance Scale (Berg) | 6 months
  Score ranging from 0 (lowest level of function) to 56 (highest level of function) with a 5-Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Gefen, Principal Investigator — ALYN Hospital Pediatric and Adolescent Rehabilitation Center
Locations (1):
- ALYN Hospital Pediatric and Adolescent Rehabilitation Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No